CLINICAL TRIAL: NCT05547529
Title: An Open-Label Randomized Clinical Trial to Evaluate the Efficacy of Neoadjuvant Chemoradiotherapy in Comparison With Neoadjuvant Chemotherapy in Patients With Resectable Squamous Cell Esophageal Cancer cT3-4aN0M0, cT1-4aN1-3M0.
Brief Title: The Efficacy of Neoadjuvant Chemoradiotherapy in Comparison With Neoadjuvant Chemotherapy in Patients With Resectable Squamous Cell Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCHENEC
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Chemoradiotherapy (Active Comparator): Carboplatin (AUC 2 mg/mL per min) and Paclitaxel (50 mg/m2 of body-surface area) were administered intravenously for five cycles, starting on days 1, 8, 15, 22, and 29. A total radiation dose of 41,4 Gy was given in 23 fractions of 1,8 Gy, 5 days per week.
  After neoadjuvant therapy, patients receive Ivor-Lewis or Mckeown Esophagectomy.
  Interventions: Procedure: Patients undergoing neoadjuvant chemoradiotherapy plus Ivory-Lewis or McKeown esophagectomy.
- Neoadjuvant Chemotherapy (Experimental): 4 cycles of DCF regimen (docetaxel 75 mg/m2 day, CDDP 75 mg/m2 and 5FU at 750 mg/m2/ day for 5 days) every 3 weeks. Patients with dysphagia 3 оr with weight loss more then 10% 6 cycles of modified-DCF regimen will be performed (mDCF, docetaxel 50 mg/m2 day, CDDP 50 mg/m2 day and 5-FU at 2400 mg/m2/day for 2 days) every 3 weeks.
  After neoadjuvant therapy, patients receive Ivor-Lewis or Mckeown Esophagectomy.
  Interventions: Procedure: Patients undergoing neoadjuvant chemotherapy plus Ivory-Lewis or McKeown esophagectomy

INTERVENTIONS:
Procedure: Patients undergoing neoadjuvant chemoradiotherapy plus Ivory-Lewis or McKeown esophagectomy. — Patients undergoing neoadjuvant chemoradiotherapy plus Ivory-Lewis or McKeown esophagectomy.
  Arms: Neoadjuvant Chemoradiotherapy
Procedure: Patients undergoing neoadjuvant chemotherapy plus Ivory-Lewis or McKeown esophagectomy — Patients undergoing neoadjuvant chemotherapy plus Ivory-Lewis or McKeown esophagectomy
  Arms: Neoadjuvant Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety, feasibility and outcomes of neoadjuvant chemotherapy followed by esophagectomy versus neoadjuvant chemoradiotherapy followed by esophagectomy for locally advanced resectable esophageal squamous cell carcinoma cT3-4aN0M0, cT1-4aN1-3M0. This is non-inferiority study (neoadjuvant chemoradiotherapy has no advantage over neoadjuvant chemotherapy).

DETAILED DESCRIPTION:
It is a prospective open-label randomized phase III clinical trial sponsored by N.N. Blokhin NMRC of Oncology. 156 patients with locally advanced resectable esophageal squamous cell carcinoma (cT3-4aN0M0, cT1-4aN1-3M0) are recruited and randomly assigned into the neoadjuvant chemoradiotherapy group (nCRT) followed by esophagectomy and the neoadjuvant chemotherapy group (nCT) followed by esophagectomy according to the proportion of 1:1. The safety, efficacy of protocols and prognosis of patients are compared between the two regimens.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histologically confirmed squamous cell carcinoma of the esophagus.
* Clinical stage cT1-4aN1-3M0 (AJCC/UICC 8th Edition).
* Indications for surgical esophageal resection
* ECOG status 0-1.
* Adequate bone marrow function (White Blood Cells > 3.0 x 109/L; Neutrophil > 2.0 × 109/L; Hemoglobin > 90 g/L; Platelets > 100 x 109/L).
* Adequate liver function (Total bilirubin < 1.5 x Upper Level of Normal (ULN); Aspartate transaminase (AST) and Alanine transaminase (ALT) < 3.0 x ULN);
* Adequate renal function (Glomerular filtration rate (CCr) > 50 ml/min.
* Adequate cardiac function. Left ventricular ejection fraction > 50%.
* Age from 18 years to 70

Exclusion Criteria:

* Clinical stage cT4bcN0cM0 (AJCC/UICC 8th Edition).
* Patients with advanced non-operable or metastatic esophageal cancer.
* Patients who have received or are receiving other chemotherapy, radiotherapy or targeted therapy.
* Patients with another previous or current malignant disease.
* Allergy or contraindications to Paclitaxel, Carboplatin, Docetaxel, Cisplatin or Fluoruracil.
* Patients with active infection of immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); HIV seropositivity; HBV DNA or HCV RNA positive.
* Severe concomitant diseases (uncontrolled arterial hypertension, diabetes mellitus, stroke less than 6 months old, mental disorders, other tumors, etc.).
* Clinically significant coronary artery disease (NYHA III / IV), congestive heart failure (NYHAIII / IV), clinically significant cardiomyopathy, myocardial infarction within the last 6 months, or high risk of uncontrolled arrhythmia.
* Chronic inflammatory diseases of the gastrointestinal tract
* Acute infectious diseases.
* Pregnancy or breast feeding.
* Serious concomitant physical and mental illness / abnormalities or territorial reasons that may prevent the patient from participating in the protocol and adherence to the protocol schedule.
* Foreigners or persons with limited legal rights.
* Any medical, geographic, or social circumstance, that in the opinion of the investigator excludes the patient's participation in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3(5) years after last patient enrolled
  Survival without local or systemic recurrence

SECONDARY OUTCOMES:
Overall survival | 3(5) years after last patient enrolled
  Overall survival of patients
Treatment related complications | During the procedure
  Сomplications after treatment
Number of cycles, frequency of neoadjuvant therapy reduction | During the procedure
  Number of chemotherapy/chemoradiotherapy cycles and doses and dose reductions
Correlation between genetic profile and tumor response | Immediately after the procedure
  Influence of the genetic profile on the tumor response
Pathological response rate(pCR) | Immediately after the surgery
  Frequency of pathological pathomorphosis
R0 resection rate | Immediately after the surgery
  Residual tumor rate

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin National Medical Research Center of Oncology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
We are not planning to share personal patient data